CLINICAL TRIAL: NCT02449239
Title: Open-Label, Multicenter, Ph 3 [Phase 3] Study to Evaluate the Efficacy and Tolerability of Intravesical Vicinium™ in Subjects With Non Muscle-Invasive Carcinoma in Situ and/or High-Grade Papillary Disease of the Bladder Treated With BCG
Brief Title: Vicinium Treatment for Subjects With Non-muscle Invasive Bladder Cancer Previously Treated With BCG
Acronym: VISTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sesen Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB4-845-02-IIIA
Record Dates: First submitted 2015-05-12; First posted 2015-05-20 (Estimated); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Bladder Cancer
Keywords: Urinary Bladder Cancer; Non-muscle invasive bladder cancer; Bladder Neoplasm; Bladder Tumor; CIS; Papillary bladder cancer; High grade bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — VB4-845

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vicinium (Experimental): Induction - 30 mg of Vicinium in 50 mL of saline administered twice weekly (BIW) for 6 weeks followed by once weekly for 6 weeks, for a total of 12 weeks.
  Maintenance - 30 mg of Vicinium in 50 mL of saline administered once weekly every other week for up to 104 weeks.
  Interventions: Biological: Vicinium

INTERVENTIONS:
Biological: Vicinium — Intravesical administration
  Other Names: VB4-845; Oportuzumab monatox

SUMMARY:
Because of the high risk for development of muscle invasive disease, cystectomy is recommended for CIS, high-grade Ta and T1 patients who experience disease recurrence following intravesical therapy. Vicinium is an experimental agent that may provide an alternative to cystectomy

DETAILED DESCRIPTION:
Bladder cancer is the 6th most common cancer in the United States, affecting more men than women. The usual first treatment for NMIBC (Ta, T1, and CIS) is transurethral resection of the bladder tumors followed by intravesical immunotherapy, most commonly with bacillus Calmette-Guérin (BCG).

Because of the high risk for development of muscle invasive disease, cystectomy is recommended for CIS and high-grade Ta and T1 patients who experience disease recurrence following intravesical therapy. For patients unable or unwilling to undergo cystectomy, treatment options are limited.

Vicinium contains the active pharmaceutical ingredient VB4-845, which is a recombinant fusion protein produced in Escherichia coli (E. coli) that expresses a humanized single-chain antibody fragment specific for the epithelial cell adhesion molecule (EpCAM) antigen linked to ETA(252-608). Once bound to the EpCAM antigen on the surface of carcinoma cells, Vicinium is internalized through an endocytic pathway. The ETA(252-608) is cleaved off and induces cell death by irreversibly blocking protein synthesis.

In vitro and in vivo pharmacology demonstrated that Vicinium exhibits potent activity [inhibitory concentration 50% (IC50) = 0.001 - 10 pM] against numerous cell lines and effectively inhibits tumor growth in several human xenograft animal models. A Phase 2 study evaluated once-weekly instillations of Vicinium 30 mg over 6 or 12 weeks, followed by up to 3 maintenance cycles (3 once-weekly instillations followed by a 9-week drug-free period) in 45 subjects with histologically-confirmed TCC of the bladder and residual CIS with or without concurrent Ta or T1 who were refractory or intolerant to BCG. A complete response (defined as no histological evidence of disease and negative urine cytology at the 3-monthly evaluations) was achieved by 44% of subjects, and 16% of subjects remained disease-free at 1-year. A post-study assessment found that these subjects were still disease-free at 18-25 months. The median time to recurrence was 134 days longer in subjects who received 12 weeks of induction therapy compared to 6 weeks.

This is an open-label, non-randomized, multicenter study in adults with NMIBC, specifically CIS (with or without papillary disease), high-grade Ta or any grade T1 papillary disease, who have previously failed BCG treatment (i.e., not those who are intolerant) with or without interferon. The study consists of a Screening period, a 12-week Induction Phase, and a Maintenance Phase of up to 21 monthly cycles for a total treatment period of up to 104 weeks. This is an outpatient study, but all treatments are administered in the study clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed non muscle-invasive urothelial carcinoma (transitional cell carcinoma) of the bladder as follows:

   1. CIS (with or without papillary disease) OR
   2. Any grade T1 papillary disease OR
   3. High-grade Ta papillary disease based on a biopsy within 8 weeks of the initial dose of study treatment. If multiple bladder biopsies are required to confirm eligibility, the last bladder biopsy to the initial dose of study treatment must be within 8 weeks. This diagnosis must be confirmed by the independent central pathology reviewer prior to subject enrollment. A subject with persistent T1 disease on the second (i.e., restaging) TURBT may be enrolled in this study only if the investigator documents the subject declines cystectomy.
2. Subjects must have received adequate BCG treatment defined as at least 2 courses of BCG, i.e., at least one induction and one maintenance course or at least 2 induction courses. The initial induction course must be at least 5 treatments within a 7-week period. The second course (induction or maintenance) must be at least 2 treatments within a 6-week period. The "5+2" doses of BCG must be given within approximately 1 year (i.e., the start of one course to start of the second course within 12 months ±1 month) and for the same disease episode for which the subject is enrolling. Treatment must be considered "full-dose" BCG (see Section 10). If additional doses or courses of BCG above the minimum "5+2" are given, these do not have to be within the same approximate 12 month timeframe.

   Subjects who were unable to receive at least 5 doses of BCG in a first course and at least 2 doses of BCG in a second course due to intolerance are not eligible.

   Subjects who began their initial course of BCG with "full-dose" BCG and required dose-reductions due to adverse events but are still able to tolerate at least "5+2" doses of BCG are considered to meet the requirement for "adequate BCG." Subjects who received less than "full dose" BCG (e.g., 1/3rd dosing) as a standard regimen and not due to dose reductions because of AEs are not eligible.

   The BCG may have been given in combination with interferon. When BCG is given simultaneously in combination with interferon, 1/3rd dosing of BCG is acceptable.
3. The subject's disease is refractory or has relapsed following adequate BCG treatment. Refractory disease is defined as disease which persists at the first evaluation following adequate BCG. Relapsed disease is defined as having a complete response to adequate BCG but recurs at a subsequent evaluation.

   Subjects will enroll into one of three cohorts based on their type of disease and the time to refractory/relapsed disease following their last dose of BCG as follows:
   * Cohort 1: Subjects with CIS with or without associated papillary disease whose disease is determined to be refractory or relapsed within 6 months of the last dose of adequate BCG treatment.
   * Cohort 2: Subjects with CIS with or without associated papillary disease whose disease is determined to be refractory or relapsed more than 6 months but within 11 months of the last dose of adequate BCG treatment.
   * Cohort 3: Subjects with high-grade Ta or any grade T1 papillary disease (without CIS) whose disease is determined to be refractory or relapsed within 6 months of the last dose of adequate BCG treatment.

   For eligibility and cohort assignment, 6 months is defined as 30 weeks i.e., 26 weeks (6 months) plus an additional 4 weeks to accommodate scheduling variations and for diagnostic work-up and 11 months is defined as 50 weeks i.e., 48 weeks (11 months) plus an additional 2 weeks to accommodate scheduling variations and for diagnostic work-up.

   For subjects enrolling in Cohort 2: The investigator documents he/she would not treat the subject with additional BCG at the time of study entry.
4. Male or non-pregnant, non-breastfeeding female, age 18 years or older at date of consent.
5. All women of childbearing potential (WOCBP) must have a negative pregnancy test within 7 days of the first dose of study therapy. A woman is not of childbearing potential if she has undergone surgical sterilization (bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy) or if she is ≥55 years of age and has had no menstrual bleeding of any kind including menstrual period, irregular bleeding, spotting, etc., for at least 12 months and there is no other cause of amenorrhea (e.g., hormonal therapy, prior chemotherapy).
6. All sexually active subjects agree to use barrier contraception (i.e., condoms) while receiving study treatment and for 120 days following their last dose of study treatment. WOCBP and males whose sexual partners are WOCBP agree to use barrier contraception and a second form of contraception while receiving study treatment and for 120 days following their last dose of study treatment.
7. Karnofsky performance status ≥ 60 (Appendix 1).
8. Adequate organ function, as defined by the following criteria:

   * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x upper limit of normal (ULN);
   * Total serum bilirubin ≤ 1.5 x ULN (CTCAE Grade ≤ 1);
   * Serum creatinine ≤ 1.5 x ULN; or a creatinine clearance ≥40 mL/min;
   * Hemoglobin ≥8.0 g/dL;
   * Absolute neutrophil count ≥1500/mm3;
   * Platelets ≥75,000/mm3
9. Ability to understand and sign an Independent Ethics Committee- or Institutional Review Board-approved informed consent document indicating that the subject (or legally acceptable representative) has been informed of all aspects of the trial and is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures. The informed consent document must be signed prior to the subject undergoing tests or procedures solely for determining study eligibility and prior to receiving any protocol treatment.

Exclusion Criteria:

1. The subject is pregnant or breastfeeding.
2. Evidence of urethral or upper tract transitional cell carcinoma (TCC) within the past 2 years. Subjects with T1 disease must have no evidence of upper or lower tract disease or a more advanced stage of disease by CT urogram or MRI urogram of the abdomen and pelvis performed within 8 weeks of the first dose of study treatment. If intravenous contrast is contraindicated, retrograde ureteropyelography, or CT or MRI without intravenous contrast may be performed.
3. Subjects with hydronephrosis, except for those subjects where hydronephrosis has been longstanding (i.e., predates the diagnosis of the CIS, Ta or T1 by more than 2 years) and diagnostic evaluation at Screening shows no evidence of tumor. Subjects with hydronephrosis that is unequivocally unrelated to upper tract malignancy may be considered eligible with Sponsor approval.
4. Any intravesicular or other chemotherapy treatment within 2 weeks or any investigational agent within 4 weeks prior to the initial dose of study drug.
5. History of recurrent severe urinary tract infections (UTIs) per investigator judgment. Subjects with a current UTI requiring antibiotic treatment may defer the initiation of Vicinium treatment on Day 1 until resolution of the UTI (even if this extends the screening period requirements to start of Vicinium treatment).
6. Active, uncontrolled impairment of the urogenital, renal, hepatobiliary, cardiovascular, gastrointestinal, neurologic or hematopoietic systems which, in the opinion of the Investigator, would predispose the subject to the development of complications from the administration of intravesical therapy and/or general anesthesia.
7. The subject has a diagnosis of another malignancy within 2 years before the first dose of study treatment, except for superficial skin cancer or localized solid tumors deemed cured by surgery and not treated with systemic anticancer therapy and not expected to require anticancer therapy in the next 2 years i.e., while the subject may be taking study treatment. However, subjects with low-risk prostate cancer, e.g.:

   * Clinically localized disease (≤T2a) and
   * Gleason score 6 (3+3) and
   * Serum PSA <10 ng/mL undergoing active surveillance may be enrolled with agreement of the sponsor.
8. A QTc interval of >470 msec by the Fridericia formula (QTcF), at the Screening ECG. If the subject's QTcF is >470 msec on the initial ECG, a total of 3 ECGs should be obtained at least 3 minutes apart and all within 30 minutes. The average of the 3 QTcF's will be used to determine eligibility. Known or suspected causes of prolonged QTc can be treated (e.g., hypocalcemia, hypokalemia, hypomagnesimia) and the ECGs may be repeated. If the subject initiates treatment with a drug known to prolong the QTc during the Screening period after the initial Screening ECGs were obtained, the Screening ECGs must be repeated once the new drug has reached steady state to ensure the average QTcF remains ≤470 msec. For subject's whose heart rate is <60 bpm, the Bazett correction formula (QTcB) may be used.
9. Subjects who, in the opinion of the Investigator, cannot tolerate intravesical administration or intravesical surgical manipulation (cystoscopy, biopsy) due to the presence of serious comorbid condition(s) (e.g., uncontrolled cardiac or respiratory disorders).
10. Local or severe allergy to any components of the drug regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-08; Primary Completion 2020-05 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minori K Rosales, M.D., Ph.D., Study Director — Sesen Bio
Locations (63):
- United States (56):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Redwood City, California
  - San Bernardino, California
  - Sherman Oaks, California
  - Torrance, California
  - Englewood, Colorado
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Daytona Beach, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Coeur d'Alene, Idaho
  - Meridian, Idaho
  - Lake Barrington, Illinois
  - Jeffersonville, Indiana
  - Fairway, Kansas
  - Lenexa, Kansas
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Glen Burnie, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Lebanon, New Hampshire
  - Brick, New Jersey
  - Lawrenceville, New Jersey
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - New York, New York
  - Poughkeepsie, New York
  - Syracuse, New York
  - The Bronx, New York
  - Concord, North Carolina
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Bryn Mawr, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Temple, Texas
  - Charlottesville, Virginia
  - Richmond, Virginia
- Canada (7):
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vicinium: Induction - 30 mg of Vicinium in 50 mL of saline administered twice weekly (BIW) for 6 weeks followed by once weekly for 6 weeks, for a total of 12 weeks.
  Maintenance - 30 mg of Vicinium in 50 mL of saline administered once weekly every other week for up to 104 weeks.
  Vicinium: Intravesical administration
Period: Induction Phase
Arm/Group | Vicinium
Started | 133
Completed | 63
Not Completed | 70
Not completed — Lack of Efficacy | 64
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1
Not completed — Patient was determined by the sponsor to be ineligible for enrollment | 1
Not completed — Withdrawal by Subject | 1
Period: Maintenance Month 3
Arm/Group | Vicinium
Started | 63
Completed | 49
Not Completed | 14
Not completed — Lack of Efficacy | 14
Period: Maintenance Month 6
Arm/Group | Vicinium
Started | 49
Completed | 36
Not Completed | 13
Not completed — Lack of Efficacy | 10
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Period: Maintenance Month 9
Arm/Group | Vicinium
Started | 36
Completed | 33
Not Completed | 3
Not completed — Lack of Efficacy | 2
Not completed — Started ibrutinib for CLL | 1
Period: Maintenance Month 12
Arm/Group | Vicinium
Started | 33
Completed | 26
Not Completed | 7
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 1
Not completed — Subject moved from area | 1
Period: Maintenance Month 15
Arm/Group | Vicinium
Started | 26
Completed | 25
Not Completed | 1
Not completed — Lack of Efficacy | 1
Period: Maintenance Month 18
Arm/Group | Vicinium
Started | 25
Completed | 25
Not Completed | 0
Period: Maintenance Month 21
Arm/Group | Vicinium
Started | 25
Completed | 23
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Sponsor decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vicinium
Number analyzed (Participants) | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 112
Age, Continuous [Mean (Full Range); unit: years] | 73.5 [54.3 to 92.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 126
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 124
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 27
  United States | 106
Disease Pathology at Enrollment [Count of Participants; unit: Participants]
  CIS with or without concomitant papillary (Ta or T1) disease | 93
  Papillary disease only | 40

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate at 3 Months
Description: Complete response rate at 3 months in patients with CIS with or without resected papillary disease following initiation of Vicinium therapy. This is the percentage of patients who were free of high-grade disease at the post-induction (3 month) assessment timepoint. A patient was considered to have a complete response if the urine cytology was reported as negative or atypical AND the cystoscopy was reported as normal or any suspicious areas were deemed negative for high-grade disease upon biopsy assessment.
Time Frame: 3 months from start of treatment
Population: Patients with CIS with or without concomitant papillary (Ta or T1) disease
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vicinium
Number analyzed (Participants) | 93
percentage of participants | 39 [29 to 49]

2. Primary Outcome: Duration of Complete Response
Description: Duration of complete response in participants with CIS with or without resected papillary disease who achieved a complete response at the post-induction (3 month) assessment. This is the number of days from the date of first occurrence of complete response to the date of documented treatment failure or death, whichever occurs first
Time Frame: Up to 24 months
Population: Participants with CIS with or without concomitant papillary (Ta or T1) disease who achieved a complete response at 3 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vicinium
Number analyzed (Participants) | 36
days | 273.0 [155.0 to NA] — The upper bound of the 95% confidence interval did not reach the 50% threshold

3. Secondary Outcome: Event-free Survival
Description: Interval from the date of first dose of study treatment to the first event (persistent high-grade disease or low grade T1 if that was the baseline disease, high-grade disease tumor recurrence, tumor progression to muscle invasive bladder cancer, cystectomy due to treatment failure, or death) prior to treatment discontinuation
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vicinium
Number analyzed (Participants) | 133
days | 90.5 [81.0 to 179.0]

4. Secondary Outcome: Complete Response Rate at 6, 9, 12, 15, 18, 21, 24 Months
Description: Complete response rate in subjects with CIS with or without resected papillary disease after 6, 9, 12, 15, 18, 21, and 24 months of Vicinium therapy. This is measured as a proportion of the total number of participants in this group that are free of high-grade disease at the respective 3-month intervals
Time Frame: Participants on treatment were assessed at months 6, 9, 12, 15,18, 21, and 24
Population: Participants with CIS with or without concomitant papillary (Ta or T1) disease
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vicinium
Number analyzed (Participants) | 93
percentage of participants
  6 months | 28 [19 to 38]
  9 months | 19 [12 to 29]
  12 months | 16 [9 to 25]
  15 months | 14 [8 to 23]
  18 months | 14 [8 to 23]
  21 months | 13 [7 to 21]
  24 months | 12 [6 to 20]

5. Secondary Outcome: Time to Cystectomy
Description: Time from the date of first dose of study treatment to physical removal of the bladder
Time Frame: Up to 48 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vicinium
Number analyzed (Participants) | 133
days | NA [NA to NA] — The median time to cystectomy was not reached due to an insufficient number of participants with events. The upper and lower limits of the 95% confidence interval could not be estimated due to an insufficient number of participants with events.

6. Secondary Outcome: Time to Disease Recurrence
Description: Time from the first dose of study treatment to the first occurrence of treatment failure or death on or prior to treatment discontinuation for participants with papillary disease only
Time Frame: Up to 24 months
Population: Participants with high-grade Ta or T1 papillary disease
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vicinium
Number analyzed (Participants) | 40
days | 436.0 [170.0 to NA] — The upper bound of the 95% confidence interval did not reach the 50% threshold

7. Secondary Outcome: Progression-free Survival
Description: Time from the date of first dose of study treatment to the date of disease progression (e.g., T2 or more advanced disease) or death on or prior to treatment discontinuation
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vicinium
Number analyzed (Participants) | 133
days | NA [NA to NA] — The median time to progression-free survival was not reached due to an insufficient number of participants with events. The upper and lower limits of the 95% confidence interval could not be estimated due to an insufficient number of participants with events.

8. Secondary Outcome: Overall Survival
Description: All participants were followed for survival during the period of consent (up to 24 months of study treatment and up to 24 months after last dose of study treatment). Any participants who were alive at last follow-up were censored.
Time Frame: Up to 48 months (up to 24 months while on study treatment and up to 24 months in the post-treatment follow-up period from the date of last dose of study drug)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vicinium
Number analyzed (Participants) | 133
days | NA [NA to NA] — The median overall survival was not reached due to an insufficient number of participants with events. The upper and lower limits of the 95% confidence interval could not be estimated due to an insufficient number of participants with events.

9. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a subject administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could, therefore, be any unfavorable and unintended sign (that may include an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. Any worsening of the participant's pre-existing medical conditions was also considered an AE, unless it was within the normal range of disease fluctuation for that participant.
Time Frame: Up to 25 months (up to 24 months of study treatment + 30 days after the last dose of study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | Vicinium
Number analyzed (Participants) | 133
Participants | 123

10. Secondary Outcome: Number of Participants That Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could, therefore, be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product, was also an adverse event. The number of participants that discontinued study treatment due to an AE was reported.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vicinium
Number analyzed (Participants) | 133
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 25 months for adverse events (up to 24 months of study treatment + 30 days after the last dose): Up to 48 months for all-cause mortality (up to 24 months of study treatment + up to 24 months of post-treatment follow-up)
Arm/Group | Vicinium
All-Cause Mortality (participants affected / at risk) | 13/133
Serious Adverse Events (participants affected / at risk) | 21/133
Other Adverse Events (participants affected / at risk) | 114/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vicinium (N=133)
Aortic valve disease (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatitis cholestasis (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (4)
Haematuria (Renal and urinary disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vicinium (N=133)
Diarrhoea (Gastrointestinal disorders) | 17 (25)
Nausea (Gastrointestinal disorders) | 16 (20)
Constipation (Gastrointestinal disorders) | 11 (18)
Abdominal pain (Gastrointestinal disorders) | 7 (12)
Vomiting (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 21 (24)
Oedema peripheral (General disorders) | 15 (16)
Pyrexia (General disorders) | 8 (10)
Urinary tract infection (Infections and infestations) | 46 (100)
Nasopharygitis (Infections and infestations) | 13 (16)
Upper respiratory tract infection (Infections and infestations) | 10 (10)
Lipase increased (Investigations) | 12 (15)
Amylase increased (Investigations) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Headache (Nervous system disorders) | 8 (9)
Dysuria (Renal and urinary disorders) | 37 (58)
Haematuria (Renal and urinary disorders) | 35 (53)
Micturition urgency (Renal and urinary disorders) | 22 (66)
Pollakiuria (Renal and urinary disorders) | 22 (54)
Urinary incontinence (Renal and urinary disorders) | 10 (11)
Bladder spasm (Renal and urinary disorders) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Hypertension (Vascular disorders) | 11 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any and all data resulting from the Study will not be presented or published in any form or media by the Institution, Investigator or Research Staff without the prior written consent of Sponsor which consent maybe as directed within the Protocol.

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT02449239/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT02449239/SAP_001.pdf